CLINICAL TRIAL: NCT05618990
Title: OPTIMIZATION of AVANCED MR SEQUENCES for BRAIN STUDIES in VOLUNTEERS (HEALTHY and PATIENTS)
Brief Title: OPTIMIZATION of ADVANCED MR SEQUENCES
Acronym: OPT-IRM
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Other Study IDs: D19-P005
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Neurosciences; MRI; Brain Tumor; Mental Disorders; Stroke
MeSH Terms: conditions — Brain Neoplasms; Mental Disorders; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This monocentric methodological study aims at optimizing advanced MR sequences for image quality (reduced artefacts, signal to noise ratio, acquisition time, stability of quantitative measurements) on a new MR unit dedicated to research in clinical and cognitive neuroscience.

DETAILED DESCRIPTION:
Primary goal : Optimization of MR protocols and validation of acquisition parameters of advanced MR sequences on healthy volunteers or patients on a new 3T MR unit dedicated to research in neurosciences.

Secondary goals

1. Perform acquisitions to validate the feasibility of research MR protocols (pilot subjects)
2. reproducibility studies

ELIGIBILITY:
Inclusion Criteria:

* 18 ans
* Covered by social security
* For women in age of procreation, under efficient contraception
* Written consent

Exclusion Criteria:

* Any MR contraindication
* Claustrophobia
* Pregnancy
* Under judiciary protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers or patients with brain lesions
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-11-05 (Actual); Primary Completion 2025-11-05 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
MR sequences optimization | 72 months
  Optimization of MR protocols and validation of acquisition parameters of advanced MR sequences on healthy volunteers or patients on a new 3T MR unit dedicated to research in neurosciences. Outcome measures depend on each pulse optimized sequence (signal-to-noise ratio, contrast-to-noise ratio, quantitative MR biomarkers).

SECONDARY OUTCOMES:
Reproducibility studies | 72 months
  Reproducibility studies (quantitative parameters, effect of denoising ...). Outcome measures depend on each pulse optimized sequence (artifacts, signal-to-noise ratio, contrast-to-noise ratio, quantitative MR biomarkers).
Pilot studies | 72 months
  Feasibility studies in cognitive neurosciences. Outcome measures depend on each MR protocol (artifacts, signal-to-noise ratio, contrast-to-noise ratio, quantitative MR biomarkers).

CONTACTS AND LOCATIONS:
Locations (1):
- OPPENHEIM Catherine, Paris, France

IPD SHARING:
Plan to Share IPD: No